CLINICAL TRIAL: NCT02023476
Title: Nerve Function in Healthy Human Volunteers With Two Different Tourniquets
Brief Title: Neurologic Examination of Wide and Narrow Tourniquets
Acronym: HEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Florian M Kovar, Univ. Lektor Dr. med. univ, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: HEM
Record Dates: First submitted 2013-12-17; First posted 2013-12-30 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Nerve Compression
MeSH Terms: conditions — Neuroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- wide tourniquet (Experimental): (Zimmer A.T.S.®3000 ) wide tourniquet MRI intervention
  Interventions: Radiation: MRI
- narrow tourniquet (Active Comparator): HemaClear ™ tourniquet MRI intervention
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — MRI- imaging on the upper arm

SUMMARY:
Nerve injury is a serious potential complication associated with the clinical use of exsanguinating tourniquets in surgery. Recently, a novel narrow tourniquet has been proposed, with the claim that it may cause less compression of the nerves. We performed an in vivo comparison of a standard wide tourniquet with the new, narrow tourniquet. Our study specifically looked at neurologic markers in the upper extremity.

DETAILED DESCRIPTION:
The HemaClear ™ OHK Medical Device HemaClear™, approved by FDA, consists of a silicon ring wrapped in a stockinet sleeve and pull straps (Fig.1). It performs three functions - blood removal (exsanguinations), arterial flow occlusion, and placement of sterile stockinet 30. The ring is placed on the extremity and then straps are pulled proximally. The silicone ring rolls up the limb while the stockinet sleeve unfolds onto the limb. During the rolling up process, the ring exerts pressure and squeezes the blood away from the limb. Application of the device takes less than a minute.

The technique behind this device is fundamentally different from classic pneumatic tourniquets, as pressure is exercised by only a single silicon ring so that the profile is very small.

Zimmer A.T.S.®3000 The A.T.S.®3000 is an automatic broad tourniquet system with a Limb Occlusion Pressure (LOP) feature. It is the latest innovation in tourniquet technology and has FDA approval. It was invented by McEwen 4 and the basic function is described in several clinical trials and publications 28. The main difference to other pneumatic tourniquets is the LOP and the Recommended tissue pressure (RTP) feature. These parameters are suitable to optimize the pressure force on the tourniquet for each individual patient. The LOP is detected before inflating the tourniquet and the RTP is the LOP plus a safety margin to guarantee a blood free field (Operator & Service Manual Zimmer A.T.S.® 3000 Automatic tourniquet system REF 60-3000-101-00).

ELIGIBILITY:
Inclusion Criteria:

* self defined Caucasian
* clinically healthy
* BMI of ≤ 30,
* a systolic arterial blood pressure ≤190 mmHg,
* no rash or dermatologic condition or tattoos which may interfere with the placement site
* no neurovascular impairment.
* all female participants received a pregnancy test at the initial screening visit.
* Study population was restricted to Caucasians to enable an assessment of device caused redness or skin lesions, not possible in a mixed study population.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Nerve compression | 20 Minutes
  mg/mm2

SECONDARY OUTCOMES:
Nerve compression | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Florian M Kovar, MD, Principal Investigator — MUW
Locations (1):
- RIAO, Sinai Hospital Baltimore, Baltimore, Maryland, United States